CLINICAL TRIAL: NCT00298051
Title: Umbilical Cord Clamping and Infant Iron Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Thrasher Research Fund (Other); Mexican National Institute of Public Health (Other Government); Instituto Mexicano del Seguro Social (Other Government); Fulbright (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 02817; 02817-8 (Other: UC Davis)
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Iron-deficiency Anemia
Keywords: Iron-deficiency anemia; Umbilical cord clamping; Infant
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Early umbilical cord clamping (control) (No Intervention): Umbilical cord was clamped immediately, or as close as possible, after delivery of the infant's shoulders. (This was standard practice in the study hospital, thus it served as the "control" group).
- Delayed umbilical cord clamping (Experimental): Umbilical cord was clamped at 2 minutes after delivery of the infant's shoulder's with the infant held at the level of the mother's uterus.
  Interventions: Procedure: Delayed umbilical cord clamping

INTERVENTIONS:
Procedure: Delayed umbilical cord clamping
  Arms: Delayed umbilical cord clamping

SUMMARY:
The aim of the study was to determine whether delayed umbilical cord clamping, as compared to early umbilical cord clamping, improves infant iron status at 6 months of age.

DETAILED DESCRIPTION:
In developing countries, up to 50% of children become anemic by 12 months of age. Risk factors for iron deficiency (ID) include low birth weight, maternal prenatal ID, and male sex. Iron deficiency anemia (IDA) during infancy and childhood is of particular concern because of the potentially detrimental effects on development, some of which may be irreversible even after treatment to correct the deficiency. Delayed umbilical cord clamping is an intervention that increases the infant's iron endowment at birth and has been shown to increase hemoglobin (Hgb) concentration at two months of age. We determined whether a two-minute delay in the clamping of the umbilical cord of normal-weight, full-term infants significantly affected infant iron and hematological status through 6 months of age. In addition, we determined whether the effect of delayed cord clamping was significantly enhanced in subgroups of infants at higher risk of developing iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women delivering at study site hospital

Exclusion Criteria:

* Delivery by Cesarean section
* Pregnancy ≤ 36 or ≥ 42 weeks gestation
* Multiple gestation
* Diagnosis of any of the following in the current pregnancy: hemorrhage requiring clinic/hospital admission, placental abnormalities, fetal anomalies, Down's syndrome of the fetus
* Diagnosis of pre-eclampsia or eclampsia in current or previous pregnancies
* Diagnosis at any time for the mother of any of the following: Diabetes, hypertension, cardiopathies, chronic renal disease
* Infant with major congenital malformation
* Infant birth weight less than 2500 g
* Mother not planning to breast feed for at least 6 months
* Mother smoked during current pregnancy
* Unwilling to return for follow-up study visits at the hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2003-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Hematologic status at 6 months of age
Iron status at 6 months of age

SECONDARY OUTCOMES:
Maternal report of clinical jaundice at 3 and 14 days of age
Newborn hematocrit at 7 hours of age
Estimated maternal bleeding at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn G Dewey, PhD, Principal Investigator — University of California, Davis; Lynnette M Neufeld, PhD, Principal Investigator — Mexican National Institute of Public Health
Locations (1):
- Hospital de Gineco Obstetrica #4 "Luis Castelazo Ayala" del Instituto Mexicano del Seguro Social, Mexico City, Mexico City, Mexico

REFERENCES:
- [Result] Chaparro CM, Neufeld LM, Tena Alavez G, Eguia-Liz Cedillo R, Dewey KG. Effect of timing of umbilical cord clamping on iron status in Mexican infants: a randomised controlled trial. Lancet. 2006 Jun 17;367(9527):1997-2004. doi: 10.1016/S0140-6736(06)68889-2. PMID 16782490
- [Result] Chaparro CM, Fornes R, Neufeld LM, Tena Alavez G, Eguia-Liz Cedillo R, Dewey KG. Early umbilical cord clamping contributes to elevated blood lead levels among infants with higher lead exposure. J Pediatr. 2007 Nov;151(5):506-12. doi: 10.1016/j.jpeds.2007.04.056. Epub 2007 Sep 17. PMID 17961694